CLINICAL TRIAL: NCT06601569
Title: Predictors of Range of Motion and Balance Abnormalities in Children Diagnosed with Cerebral Palsy
Status: Recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed fekry ibrahim salman, assistant professor physical therapy department, Cairo University
Other Study IDs: P.T.REC/012/005209
Record Dates: First submitted 2024-07-27; First posted 2024-09-19 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy | interventions — Range of Motion, Articular

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- diplegic cerebral palsy
  Interventions: Diagnostic Test: balance and range of motion
- quadripledic cerebral palsy
  Interventions: Diagnostic Test: balance and range of motion
- hemiplegic cerebral palsy
  Interventions: Diagnostic Test: balance and range of motion
- dyskinetic cerebral palsy
  Interventions: Diagnostic Test: balance and range of motion

INTERVENTIONS:
Diagnostic Test: balance and range of motion — * Spinal alignment and range of motion measure scale (SAROMM): is a measure of spinal alignment and range of motion using standard physical therapy techniques scored on a 5-point ordinal score of 0 (normal alignment and range with active correction) to4 ("severe" ﬁxed deformity) (Bartlett ey al., 2005)
  * Modified Ashworth scale (MAS): is a measure of muscle motion and scoring the perceived resistance to movement on a scale of 1 (no increase in tone) to 5 (rigid in ﬂexion or extension) (Clopton et al., 2005).
  * Early clinical assessment of balance (ECAB) scale: Is a 13-item test that estimates postural stability for children with CP across all levels of functional ability (Jeffries etal., 2016).
  * Functional strength assessment scale: Therapists completed a functional strength assessment (FSA) to obtain an estimate of strength for major muscle groups including the neck and trunk ﬂexors and extensors, and hip extensors, knee extensors, and shoulder ﬂexors bilaterally.
  Other Names: Spinal alignment and range of motion measure scale; Modified Ashworth scale (MAS); Early clinical assessment of balance (ECAB) scale; Functional strength assessment scale

SUMMARY:
1. To better understand the factors that contribute to ROM abnormalities in children diagnosed with CP.
2. To describe the distribution of primary (muscle tone and postural stability)and secondary impairments (ROM and functional muscle strength) across the gross motor spectrum measured by GMFCS scores.
3. To evaluate the effects of primary and secondary impairments on gross functional outcome in children with spastic CP.
4. To find any possible correlation between clinical variables.

ELIGIBILITY:
Inclusion Criteria:

* only children with clinical diagnosis of cerebral palsy , who were receiving physiotherapy services at the paediatric out-patient clinic of Faculty of Physical Therapy, Cairo University for a minimum of six months regularly.

Exclusion Criteria:

* Children were excluded if they had one or more of the following: behavioral issues, a history of persistent heart or chest disease, significant visual or auditory impairment, botulinum toxin injection at last six months prior to the study.

Ages: 18 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: children with cerebral plasy their age ranged fro 18 month t 5 yeas old
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
predictors of range of motion and balance abnormalities | from 1 august 2024 to 1 october 2024
  the aim of the study is to investigate the predicted cause if the range of motion abnormalities measured by (spinal alignment and range of motion assessment scale ) and balance abnormalities ( measured by early clinical assessment of balance scale )in children with cerebral palsy like muscle strength (measured by functional muscle strength scale) and muscle tone changes (measured by modified athwart scale)

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physical Therapy Cairo University, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes